CLINICAL TRIAL: NCT06449989
Title: Comparison of Molecular-Genetic Concordance of the Primary Tumor and Brain Metastases of Colorectal Cancer
Acronym: GENCONCOR-1
Status: Recruiting | Type: Observational
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, David Halafyan, Physician-researcher, Blokhin's Russian Cancer Research Center
Other Study IDs: 115522143966
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer Metastatic; Brain Metastases, Adult; Ras (KRAS or NRAS) Gene Mutation; BRAF Gene Mutation; HER2 Gene Mutation; MSI
Keywords: Colorectal Cancer Metastatic; Brain Metastases, Adult; Ras (KRAS or NRAS) Gene Mutation; BRAF Gene Mutation; HER2 Gene Mutation; MSI
MeSH Terms: conditions — Brain Neoplasms | interventions — Genes, mos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival formalin-fixed and paraffin-embedded tumor blocks (pair of matched tumor samples: from the primary tumor and from intracranial metastases)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Tumor samples will be tested for mutation status of KRAS, NRAS, BRAF, HER2 and MSI — For molecular genetic research, archival formalin-fixed and paraffin-embedded tumor blocks will be used. Research method - HRM-PCR sequencing to determine mutation status of KRAS, NRAS and BRAF (RotorGene 6000, ABI Prism 3500) and fragmentation analysis to determine MSI (ABI Prism 3500) Subject to study: mutations in the KRAS, NRAS, BRAF genes, as well as MSI status and HER2neu expression (± amplification) Somatic mutations in the RAS family genes are planned to be studied in exons 2 (codons 12 and 13), exon 3 (codon 61) and exon 4 (codon 146). In the case of the BRAF gene - exon 15 (codons 597-601). Determination of microsatellite instability is planned using five markers: BAT25, BAT26, NR21, NR24, NR27, associated with structural and functional disorders of the DNA unpaired base repair system.
  Assessment of HER2 gene status is planned by immunohistochemical (IHC) screening of HER2neu expression. IHC-screening of HER2-status will be performed using an antibody clone 4B5 (Ventana).

SUMMARY:
GENCONCOR-1 study is translational research aimed to investigate the concordance of the molecular genetic profile of the primary tumor and brain metastases (BM) of colorectal cancer (CRC). The study was conducted by post hoc analysis of pairs of samples of histological material with determination of the mutational status of genes KRAS, NRAS, BRAF, HER2 and MSI.

DETAILED DESCRIPTION:
Brain metastases (BM) from colorectal cancer (CRC) are a rare event reported in less than 3% of patients with CRC (the reported incidence ranges from 0.27 to 3%). This course is associated with a poor prognosis. Treatment of these patients remains challenging. Nevertheless, given the rarity of the event, at this time not enough is known about molecular biology of BM from colorectal cancer and its concordance with matched primary tumors.

In N.N. Blokhin National Medical Research Center of Oncology over 26 years (1998-2024) identified 108 patients with BM from CRC. Of this number, 72 patients had a history of neurosurgical resection of BM. In turn, for 32 patients access to a pair of tumor samples: from the primary tumor and from intracranial metastases. Tumor samples will be tested for mutation status of genes KRAS, NRAS, BRAF, HER2 and MSI. Analysis was limited to this pool of genes because of their clinical relevance and potential prognostic information. The molecular profile of the BM will be compared with the corresponding primary tumor with calculation of concordance rate (%).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Histologically confirmed cancer of the colon or rectum.
3. Histologically confirmed metastatic lesion of the brain.
4. Neurosurgical resection for brain metastases of colorectal cancer.
5. Presence of paired tumor samples (both primary tumor and intracranial material).

Exclusion Criteria:

1. Missing one sample from a pair of tumor samples.
2. Low quality or lack of tumor material for molecular genetic research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer (CRC) and brain metastases (BM) will be analyzed according to sex, age, functional status (ECOG 0-1 or 2-3), number of BM (solitary or ≥ 2), clinical manifestations of BM (symptomatic or asymptomatic), extracranial lesions at the time of diagnosis BM (present or absent), course of brain metastases (synchronous with the primary tumor or metachronous), side of the location of the primary tumor (left-sided or right-sided CRC), location of intracranial lesions (supratentorial or subtentorial), number of previous lines of drug therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Concordance rate (%) | 1 month
  Concordance rate (%) between mutational status of the brain lesions and their corresponding primary tumor. Calculated as the ratio of concordant cases to total cases.

SECONDARY OUTCOMES:
Intracranial progression-free survival (CNS-PFS1) | 3 months
  Time from the date of cancer diagnosis to the date of detection of brain metastases.
Overall survival (OS) | 6 months
  Time from the date of detection of brain metastases to the date of death.
Intracranial progression-free survival (CNS-PFS2) | 3 months
  Time from the date of neurosurgical resection to the date of intracranial progression (continued growth or distant brain metastases) or death.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Tryakin, MD, professor, Study Chair — Blokhin's Russian Cancer Research Center; Ali Bekyashev, MD, professor, Study Chair — Blokhin's Russian Cancer Research Center; Anna Stroganova, MD, Study Chair — Blokhin's Russian Cancer Research Center
Locations (1):
- Blokhin's Russian Cancer Research Center, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in article, after deidentification (text, tables, figures, and appendices)
Time Frame: From the moment of publication of the results and indefinitely
Access Criteria: For individual participant data meta-analysis. Data will be available indefinitely in the appendix of the published article